CLINICAL TRIAL: NCT07325344
Title: Active Locomotion of Magnetically Controlled Capsule Endoscopy With Small Bowel Insufflation or Water Infusion: A Feasibility Study
Brief Title: Active Locomotion of Magnetically Controlled Capsule Endoscopy in the Small Bowel: A Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of Gastroenterology Department, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KYLL-2025-10-008-1
Record Dates: First submitted 2025-12-16; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Capsule Endoscopy
Keywords: capsule endoscopy; small bowel disease; locomotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subject (Experimental): During the routine air/water insufflation phases of the enteroscopy, the researchers will attempt to guide the capsule's movement using an external magnetic control device.
  Interventions: Device: magnetic control

INTERVENTIONS:
Device: magnetic control — Intervention: On the day of the examination, the subject will swallow the capsule endoscope. This will be followed by a standard enteroscopy procedure. During the routine air/water insufflation phases of the enteroscopy, the researchers will attempt to guide the capsule's movement using an external magnetic control device.

SUMMARY:
The aim of this study is to evaluate the responsiveness of the capsule endoscope to the attitude controller and to investigate its active locomotion performance within the small bowel.

DETAILED DESCRIPTION:
During the standard air insufflation or water infusion phases of double-balloon enteroscopy, researchers will use a handheld controller to try to steer the capsule. At the same time, the real-time imaging from both the enteroscope and the capsule will be simultaneously monitored to assess the capsule's active movement and its responsiveness to control.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo enteroscopy.

Exclusion Criteria:

* Patients with severe dysfunction of vital organs (e.g., heart, lungs). Patients with small bowel obstruction precluding adequate bowel preparation. Patients with a history of multiple abdominal surgeries. Patients with implanted devices such as cardiac pacemakers or metal implants. Patients with other high-risk conditions or lesions (e.g., moderate-to-severe esophagogastric varices, massive ascites).

Patients who are pregnant or lactating. Patients unable or unwilling to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
capsule endoscope's responsiveness to the attitude controller | During performing double-balloon enteroscope
  Excellent: The magnetically controlled capsule endoscope can precisely follow the attitude controller to move to the target area.
  Moderate: The magnetically controlled capsule endoscope can follow the attitude controller's movement, but cannot be accurately guided to the target area.
  Poor: There are signs of magnetic attraction, but the capsule does not follow the movement of the attitude controller.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China